CLINICAL TRIAL: NCT01504347
Title: Randomized, Double-Blind, Phase 1/2 Clinical Study to Investigate the Safety and Immunogenicity of a Multivalent Recombinant OspA Lyme Borreliosis Vaccine (mv rOspA LB Vaccine) in Healthy Subjects Aged 18 to 70 Years
Brief Title: Phase 1/2 Lyme Vaccine Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxter Innovations GmbH (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 730901; 2010-023384-18 (EudraCT Number)
Record Dates: First submitted 2011-12-22; First posted 2012-01-05 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Prophylaxis of Lyme Borreliosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Primary vaccination in seronegative subjects (Experimental)
  Interventions: Biological: Multivalent recombinant OspA Lyme Borreliosis Vaccine
- Booster vaccination in seronegative subjects (Experimental)
  Interventions: Biological: Multivalent recombinant OspA Lyme Borreliosis Vaccine
- Primary + booster vacc. (seronegative + seropositive subjects) (Experimental)
  Interventions: Biological: Multivalent recombinant OspA Lyme Borreliosis Vaccine

INTERVENTIONS:
Biological: Multivalent recombinant OspA Lyme Borreliosis Vaccine — Primary vaccination (6 study arms of 50 subjects each): 3 intramuscular injections containing either dose A, B or C in an adjuvanted or non-adjuvanted formulation (6 different formulations) given in monthly intervals (recruited in 3 sequential cohorts)
  Arms: Primary vaccination in seronegative subjects
Biological: Multivalent recombinant OspA Lyme Borreliosis Vaccine — Booster vaccination 9-12 months after first vaccination in Section 1 subjects
  Arms: Booster vaccination in seronegative subjects
Biological: Multivalent recombinant OspA Lyme Borreliosis Vaccine — 3 intramuscular injections at monthly intervals (using 2 formulations selected from Section 1) in seronegative and seropositive subjects (N=350) and a booster vaccination at 6 months or at 9-12 months (Cohorts 4: seronegatives; Cohort 5: seropositives)
  Arms: Primary + booster vacc. (seronegative + seropositive subjects)

SUMMARY:
Section 1:

The purpose of the study is to obtain safety and immunogenicity data of different dose levels of a multivalent recombinant OspA Lyme Borreliosis (mv rOspA LB) Vaccine with and without adjuvant in seronegative healthy adults aged 18 to 70 years. The outcome shall provide the basis for dose/formulation selection for Section 2 of the study.

Section 2:

An additional purpose of the study is to evaluate the safety and immunogenicity of the optimal dose(s)/formulation of the mv rOspA LB Vaccine in a larger population of seronegative and seropositive healthy subjects aged 18 to 70 years.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject is 18 to 70 years old at the time of screening
* Subject has an understanding of the study, agrees to its provisions, and gives written informed consent prior to study entry
* Subject is generally healthy, as determined by the investigator's clinical judgment through collection of medical history and the performance of a physical examination
* If female of childbearing potential, presents with a negative urine pregnancy test, and agrees to employ adequate birth control measures for the duration of the study

Additional inclusion criterion for seropositive subjects in Section 2 only:

- Subject is seropositive for Borrelia burgdorferi sensu lato (s.l.) antibodies at study entry

Main Exclusion Criteria:

* Subject has a physician-diagnosed chronic illness related to Lyme borreliosis (LB) or active LB
* Subject has been treated for LB with antibiotics within 3 months of study entry
* Subject had a tick bite within 3 weeks prior to screening or first vaccination
* Subject has a history or active infection with Babesia microti (babesiosis) or Anaplasma phagocytophilum (ehrlichiosis)
* Subject currently has or has a history of significant cardiovascular, respiratory (including asthma), metabolic, neurological, hepatic, rheumatic, autoimmune, hematological, gastrointestinal or renal disorder
* Subject has clinically significant abnormal laboratory values at screening
* Subject currently has or has a history of immunodeficiency
* Subject tests positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV)
* Subject has a disease or is currently undergoing a form of treatment or was undergoing a form of treatment within 30 days prior to study entry that could be expected to influence immune response.
* Subject has a history of anaphylaxis or severe allergic reactions
* Subject has received any live vaccine within 4 weeks or inactivated vaccine within 2 weeks prior to vaccination in this study
* Subject is pregnant or lactating at the time of study enrollment

Additional exclusion criterion for subjects in Section 1 and seronegative subjects in Section 2:

- Subject is seropositive for Borrelia burgdorferi sensu lato (s.l.) antibodies at study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1630 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2011-09-13 (Actual); Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
Antibody response to the vaccine | 28 days after the third vaccination (= Day 85)
Frequency and severity of injection site and systemic reactions | Within 7 days after each vaccination (i.e. Days 8, 36 and 64)

SECONDARY OUTCOMES:
Antibody response | At baseline, 28 days after each vaccination (i.e. Days 29, 57 and 85), 180 and 270 days after the first vaccination (Day 181, Day 271) and 180 days after the booster vaccination (Day 361 or Day 451 - 546)
Fold increase in antibody titer compared to baseline | 28 days after each vaccination, 180 and 270 days after the first vaccination and 180 days after the booster vaccination
Seroconversion rate (at least 4-fold increase of each rOspA type-specific Immunoglobulin G (IgG) titer) as compared to baseline | 28 days after each vaccination, 180 and 270 days after the first vaccination and 180 days after the booster vaccination
Frequency and severity of adverse events | 28 days after each vaccination and during entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- Austria (2):
  - Medical University Vienna, Dept. of Clinical Pharmacology, Vienna
  - Zentrum für Reisemedizin (Center for Travel Medicine), Vienna
- Germany (6):
  - Berliner Centrum für Reise- und Tropenmedizin GmbH (BCRT), Berlin
  - GWT-TUD GmbH, Dresden
  - Hautarztpraxis Cutanis (Dermatologist), Freiburg im Breisgau
  - Internistische Gemeinschaftspraxis (Internal Medicine Group Practice), Mainz
  - Innomed Dr. Naudts Klinische Forschung, Rodgau
  - Universitätsklinikum Tübingen, Abtlg. Tropenmedizin, Tübingen

REFERENCES:
- [Derived] Wressnigg N, Barrett PN, Pollabauer EM, O'Rourke M, Portsmouth D, Schwendinger MG, Crowe BA, Livey I, Dvorak T, Schmitt B, Zeitlinger M, Kollaritsch H, Esen M, Kremsner PG, Jelinek T, Aschoff R, Weisser R, Naudts IF, Aichinger G. A Novel multivalent OspA vaccine against Lyme borreliosis is safe and immunogenic in an adult population previously infected with Borrelia burgdorferi sensu lato. Clin Vaccine Immunol. 2014 Nov;21(11):1490-9. doi: 10.1128/CVI.00406-14. Epub 2014 Sep 3. PMID 25185574
- [Derived] Wressnigg N, Pollabauer EM, Aichinger G, Portsmouth D, Low-Baselli A, Fritsch S, Livey I, Crowe BA, Schwendinger M, Bruhl P, Pilz A, Dvorak T, Singer J, Firth C, Luft B, Schmitt B, Zeitlinger M, Muller M, Kollaritsch H, Paulke-Korinek M, Esen M, Kremsner PG, Ehrlich HJ, Barrett PN. Safety and immunogenicity of a novel multivalent OspA vaccine against Lyme borreliosis in healthy adults: a double-blind, randomised, dose-escalation phase 1/2 trial. Lancet Infect Dis. 2013 Aug;13(8):680-9. doi: 10.1016/S1473-3099(13)70110-5. Epub 2013 May 10. PMID 23665341